CLINICAL TRIAL: NCT04524923
Title: Touch Screen Usage Time In Relation To Visual Motor Integration and Quality of Life In Preschoolers: A Cross Sectional Study
Brief Title: Touch Screen Usage Time In Relation To Visual Motor Integration and Quality of Life In Preschoolers
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira M Abd-elmonem, PHD, principle investigator, Cairo University
Other Study IDs: child development
Record Dates: First submitted 2020-08-21; First posted 2020-08-24 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Child Development
Keywords: Cognitive development; Digital devices; Quality of Life Inventory; Visual motor integration; touch screen usage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cohort group: Ninety-seven typically developing preschool children of both genders with age ranges from three to five years will be included in this study. Visual motor integration, quality of life and cognitive function were assessed by the Peabody Developmental Motor Scale, the Pediatric Quality of Life Inventory™ and the Pediatric Quality of Life Inventory™ cognitive functioning scale respectively
  Interventions: Other: visual motor integration; Other: Quality of life assessment; Other: Cognitive Functioning

INTERVENTIONS:
Other: visual motor integration — investigate the relation between touch screen usage and visual motor integration in preschoolers
Other: Quality of life assessment — investigate the relation between touch screen usage and Quality of life assessment in preschoolers
Other: Cognitive Functioning — investigate the relation between touch screen usage and Cognitive Functioning assessment in preschoolers

SUMMARY:
Recent literatures are associating digital technology extensive and addictive use with physical, psychosocial and cognitive inverse consequences. This research focuses more on number of touch screen devices; age started using devices and usage time in relation to cognitive function in preschoolers.

DETAILED DESCRIPTION:
A hundred typically developing preschool children of both genders with age ranges from three to five years will be included in this study. Visual motor integration, quality of life and cognitive function were assessed by the Peabody Developmental Motor Scale, the Pediatric Quality of Life Inventory™ and the Pediatric Quality of Life Inventory™ cognitive functioning scale respectively

Sample size To avoid type II error, sample size calculation was based on data from a pilot study on correlation between touch screen usage time and visual motor integration. Using G*POWER statistica software (version 3.1.9.2; Franz Faul, Universitat Kiel, Germany) [Correlational study, α=0.05, β=0.2, and medium effect size = 0.3] revealed that the appropriate sample size for this study was N=84 Therefore, one-hundred children were recruited for possible dropouts during assessment.

ELIGIBILITY:
Inclusion criteria:

Children were enrolled in this study according to the following criteria:

* Age ranges from three to five years.
* Both genders were included.

Exclusion criteria:

Children were excluded from the study if they had any of the following criteria:

* Diagnosed with attention deficit/hyperactivity disorder (ADD/ADHD) or developmental co-ordination disorder (DCD).
* Preterm children; children with major physical disabilities, genetic disorders; prenatal exposure to alcohol; children with a history of head trauma and infections.
* Diagnosed with psychiatric conditions such as autism and depression.
* Diagnosed with significant behavioral disorders
* Diagnosed with fine motor problems.
* Significant auditory or visual deficits.

Ages: 3 Years to 5 Years | Sex: All
Age Groups: Child
Study Population: This study will be delimited to typically developing preschool children, from both genders, with age ranging from three to five years.
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
visual motor integration | 1 September 2020 to 31 March 2021
  The Peabody Developmental Motor Scale will be used to assess visual motor integration. It is a standardized, norm-referenced test used for the assessment of upper limb functions. It is an early childhood motor development program that provides (in one package) both in depth assessment and training of gross and fine motor skills. It can be used by occupational therapists, physical therapists, psychologists, and others who are interested in examining the motor abilities of young children. It is composed of six subtests:-Reflexes (8 items), stationary (30 items), locomotion (89 items), object manipulation (24 items), grasping (25 items) and visual motor integration (72 items). The results of the subtests may be used to generate 3 global indexes of motor performance called (composites). These composites are gross motor quotient, fine motor quotient and total motor quotient with higher scores represent better performance
Physical and Psychosocial Health | 1 September 2020 to 31 March 2021
  The Pediatric quality of life inventory™ generic Arabic parent proxy-report for children from two to five years was used to assess quality of life. It was developed to quantify health- related quality of life (HRQoL) of children and adolescents aged 2-18 years. It consists of 23 questions and evaluate how frequently of a trouble the child has had over the past month. Interpretation of the scale reveals the mean performance as total scale score, physical functioning score (eight questions), emotional functioning score (five questions), social functioning score (five questions) and school function scores (five items). the scores are from 0 to 100 with higher results reflecting better performance.
cognitive function | 1 September 2020 to 31 March 2021
  Pediatric Quality of Life Inventory™ Cognitive Functioning Scale will be used to assess cognitive function. It was developed as a brief generic symptom-specific instrument to measure cognitive functioning. The 6-item scale was designed as a brief and easy-to-administer patient self-reported and parent proxy-reported generic symptom specific instrument to measure cognitive functioning across pediatric populations, originally developed in a pediatric cancer population. The PedsQLTM Cognitive Functioning Scale includes format, instructions, Likert scale from 0 to 100 with higher scores indicating better cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Amira M El-tohamy, Phd, Study Chair — Cairo University; Amira M Mahmoud, Study Director — Cairo University
Locations (1):
- faculty of physical therapy, Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No